CLINICAL TRIAL: NCT00171054
Title: A Randomized, Double-blind, Parallel Group, Active-controlled, 38-week Study to Evaluate the Efficacy of Valsartan Versus Amlodipine on the Arterial Properties of Postmenopausal Women With Mild to Moderate Hypertension
Brief Title: Efficacy and Safety of Valsartan Versus Amlodipine in Postmenopausal Women With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAL489A2418
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: hypertension; postmenopausal; valsartan; amlodipine; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Valsartan 320 mg (Experimental)
  Interventions: Drug: Valsartan 320 mg; Drug: Hydrochlorothiazide
- Amlodipine 10 mg (Experimental)
  Interventions: Drug: Amlodipine 10 mg; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan 320 mg — Patients received 160 mg valsartan for 4 weeks. Patients were then up-titrated to receive either 320 mg valsartan for the following 8 weeks.
  Arms: Valsartan 320 mg
Drug: Amlodipine 10 mg — Patients received 5 mg amlodipine for four weeks. Patients were then up-titrated to receive 10 mg amlodipine for the following 8 weeks.
  Arms: Amlodipine 10 mg
Drug: Hydrochlorothiazide — At Week 12, patients who did not meet target Blood Pressure for both Systolic Blood Pressure < 140 mmHg and Diastolic Blood Pressure < 90 mmHg were eligible to receive 12.5 mg open-label Hydrochlorothiazide for the following 26 weeks.

SUMMARY:
The purpose of this study is compare treatment with valsartan with the possible addition of a diuretic, hydrochlorothiazide, on high blood pressure with the drug amlodipine with the possible addition of a diuretic, hydrochlorothiazide. In particular, the effect of treatment on the stiffness of the blood vessels will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Mild to moderate hypertension
* Statin therapy or LDL≤ 4.1 mmol/L

Exclusion Criteria:

* Severe hypertension
* LDL > 4.1 mmol/L if not taking anti-hyperlipidemic medication
* Certain hormonal therapy
* History of stroke, myocardial infarction, heart failure, chest pain, abnormal heart rhythm
* Liver, kidney, or pancreas disease
* Diabetes
* Raynaud's disease or any other significant peripheral vascular disease
* Allergy to certain medications used to treat high blood pressure

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2003-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Valsartan 320 mg: Double-blind study medication consisted of valsartan 160 mg capsules for oral administration. Open-label HCTZ 12.5 mg (orally administered) was electively prescribed at week 12.
- Amlodipine 10 mg: Amlodipine, orally administered, was provided as 5 mg capsules. Open-label HCTZ 12.5 mg (orally administered) was electively prescribed at week 12.
Period: Overall Study
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Started | 63 | 62
Completed | 53 | 50
Not Completed | 10 | 12
Not completed — Protocol Violation | 1 | 2
Not completed — Patient withdrew consent | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 8 | 8
Not completed — Condition no longer required study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg | Total
Number analyzed (Participants) | 63 | 62 | 125
Age Continuous [Mean (Standard Deviation); unit: years] | 62.3 (5.76) | 60.4 (5.08) | 61.4 (5.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 62 | 125
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 38 in the Carotid-femoral Pulse Wave Velocity (PWV)
Description: PWV was determined from transcutaneous Doppler flow recordings and the foot-to-foot method triggered by the simultaneous ECG. Two simultaneous Doppler flow tracings were taken at the left common carotid and the right femoral artery in the groin with a linear array probe. The time delay (t) was measured between R wave of the ECG and the base of the flow waves recorded at these points, and averaged over 10 beats. The distance (D) traveled by the pulse wave was measured over body surface as the distance from the suprasternal notch to the carotid artery. PWV was calculated as PWV=D/t.
Time Frame: Baseline and Week 38
Population: Intent-to-treat. The intent to treat population is defined as those who provide a baseline measure and at least one post-baseline measurement (not necessarily an endpoint measure)
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 56 | 53
m/s | -1.9 (0.29) | -1.7 (0.30)

2. Secondary Outcome: Change From Baseline in Post-ischemic Forearm Skin Reactive Hyperemia at Week 12
Description: Cutaneous blood flow was continuously recorded by a laser Doppler flowmeter. The laser Doppler flow probe was applied on the volar part of the right forearm with a plastic holder 10 cm proximal to the wrist. All measurements were made with a pressure cuff on the arm and inflated 20 mmHg above systolic BP and maintained for 2 min then rapidly deflated. All measurements were made in a quiet room with a patient in the supine position. The maximal reactive hyperemia was measured after cuff deflation, which allows measurement of the right forearm postischemic skin reactive hyperemia (SRH).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Perfusion units
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 54 | 53
Perfusion units | 25.4 (14.88) | -105.6 (15.31)

3. Secondary Outcome: Change From Baseline in Post-ischemic Forearm Skin Reactive Hyperemia at Endpoint (Week 38)
Description: as for outcome 2
Time Frame: Week 38
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Perfusion units
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 55 | 53
Perfusion units | -9.7 (13.73) | -94.6 (14.20)

4. Secondary Outcome: Change From Baseline for Endothelial Function Measured by Brachial Artery Flow-mediated Vasodilatation (FMD) Using the Brachial Artery Reactivity Test (BART) at Week 12
Description: Endothelial function will be assessed using high-resolution duplex ultrasound with wall tracking to measure FMD of the brachial artery during reactive hyperemia. FMD of the brachial artery in response to reactive hyperemia in the distal forearm (and glyceryl trinitrate as a non-endothelium dependent control) will be measured from B-mode ultrasound images using a standard 7 MHz linear array transducer and HDI 5000 system with edge detection.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 56 | 49
percent | -8.7 (0.35) | -8.6 (0.38)

5. Secondary Outcome: Change From Baseline for Endothelial Function Measured by Brachial Artery Flow-mediated Vasodilatation (FMD) Using the Brachial Artery Reactivity Test (BART) at End-point (Week 38)
Description: as for outcome 4
Time Frame: Baseline and Week 38
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 56 | 51
percent | -8.1 (0.53) | -8.2 (0.56)

6. Secondary Outcome: Changes in Mean Left Carotid Distensibility at Week 12
Description: For carotid distensibility, the left and right bulbs and common carotid arteries are measured using tissue Doppler imaging with the linear array probe. Absolute diameter and diameter changes over the cardiac cycles will be recorded. Distensibility of each bulb will be calculated for three consecutive heart cycles and averaged and corrected for blood pressure.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 54 | 51
percent | 0.0 (0.14) | 0.0 (0.15)

7. Secondary Outcome: Changes in Mean Left Carotid Distensibility at Week 38
Description: as for outcome 6
Time Frame: Baseline and Week 38
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 54 | 53
percent | 0.0 (0.16) | 0.1 (0.16)

8. Secondary Outcome: Changes in Mean Right Carotid Distensibility at Week 12
Description: as for outcome 6
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 54 | 52
percent | -0.4 (0.16) | 0.1 (0.17)

9. Secondary Outcome: Changes in Mean Right Carotid Distensibility at Week 38
Description: as for outcome 6
Time Frame: Baseline and Week 38
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 54 | 53
percent | -0.2 (0.17) | 0.0 (0.17)

10. Secondary Outcome: Changes in Baroreflex Sensitivity as it Relates to Changes in Carotid Distensibility From Baseline to Week 12
Description: The calculation of spontaneous baroflex sensitivity was obtained by the sequence method. Baroflex sequences are defined by at least three consecutive beats in which the systolic blood pressure and the RR interval of the following beat either both increased or decreased. The slope of each individual sequence is computed and the mean slope is determined as the average of all slopes within a given period of time and taken as the gain of the cardiac baroflex (BRSs).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: EP
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 55 | 52
EP | 1.5 (1.71) | -1.5 (1.78)

11. Secondary Outcome: Changes in Baroreflex Sensitivity as it Relates to Changes in Carotid Distensibility From Baseline to Week 38
Description: as for outcome 10
Time Frame: Baseline and Week 38
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: EP
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 56 | 52
EP | -2.0 (1.38) | 0.1 (1.44)

12. Secondary Outcome: Change in Left Ventricular Mass Index (LVMI) and Diastolic Function Using Echocardiography From Baseline to Week 38
Time Frame: Baseline and Week 38
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 19 | 22
percent | -4.8 (2.43) | -6.2 (2.13)

13. Secondary Outcome: Changes in Central Blood Pressure, Evaluated by Applanation Tonometry From Baseline at Weeks 12 and 38
Description: Central Blood Pressure was measured via applanation tonometry recordings of the common carotid artery and from brachial oscillometric recordings. The Simultaneously obtained carotid artery pressure and standard brachial artery blood pressure are computed to obtain the central systolic pressure.
Time Frame: Baseline, Week 12 and Week 38
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Number analyzed (Participants) | 56 | 53
mm Hg
  Week 12 | -9.1 (1.06) | -14.2 (1.10)
  Week 36 | -11.1 (1.07) | -13.9 (1.12)

ADVERSE EVENTS:
Arm/Group | Valsartan 320 mg | Amlodipine 10 mg
Serious Adverse Events (participants affected / at risk) | 2/63 | 2/62
Other Adverse Events (participants affected / at risk) | 35/63 | 51/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 320 mg (N=63) | Amlodipine 10 mg (N=62)
Diplopia (Eye disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 320 mg (N=63) | Amlodipine 10 mg (N=62)
Vertigo (Ear and labyrinth disorders) | 4 | 2
Asthenia (General disorders) | 5 | 2
Fatigue (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 9 | 48
Bronchitis (Infections and infestations) | 8 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache (Nervous system disorders) | 6 | 5
Insomnia (Psychiatric disorders) | 4 | 1
Hypotension (Vascular disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.